CLINICAL TRIAL: NCT03561181
Title: A Single-center, Open, Phase I Clinical Trial to Evaluate Safety of S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine in Healthy Volunteers Aged Above 3 Months
Brief Title: Safety Study of S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine in Healthy Volunteers Aged Above 3 Months
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201619306
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Dysentery; Dysentery, Bacillary
MeSH Terms: conditions — Dysentery; Dysentery, Bacillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose Group (Experimental): Received Vaccine: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine,10μg/dose
  Interventions: Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine
- low dose Group (Experimental): Received Vaccine: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine,5μg/dose
  Interventions: Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine

INTERVENTIONS:
Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine — Group 1:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 10 µg S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine.
  Arms: High dose Group
Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine — Group 2:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 5 µg S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine.
  Arms: low dose Group

SUMMARY:
The purpose of this study is to evaluate safety of S.flexneriza-S.sonnei Bivalent Conjugate Vaccine in healthy volunteers aged above 3 Months.

ELIGIBILITY:
Inclusion Criteria:

* 3 months old and above healthy people.
* Subject or legal representative who consent and has signed written informed consent.
* Subject and parent/guardian who is able to comply with all study procedures.
* Subject who did't receive blood products within 30 days ,immune with any live vaccine within 14 days and inactivated vaccine within 7 days before vaccination.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* Febrile illness (temperature ≥ 38°C) in the 3 days.
* Subject who are allergic to tetanus toxoid.
* Allergic history after vaccination.
* Immunodeficiency diseases patients who administered with immunosuppressive agents.
* In pregnancy or lactation or pregnant women.
* Subject who are suffering from serious chronic diseases, infectious diseases, active infection, cardiovascular disease,liver or kidney disease.
* Subject who have symptoms such as diarrhea, abdominal pain, and pus and bloody stools in the past 3 days.
* History of allergy，eclampsia, epilepsy,brain trauma,encephalopathy and mental disease or family disease.
* Subject who diagnosis of thrombocytopenia or other history of coagulopathy may cause intramuscular contraindication.
* Children with abnormal labor（pregnancy week<37w,>42w）,birth weight (<2500g,>4000g), asphyxia rescue history,congenital malformations or developmental disorders(Only applicable to 3-5 months old group)
* Blood routine, blood chemistry and urinalysis laboratory collection abnormalities and the severity of grade 2 and above before immunization.
* Subject who plan to participate in or is in any other drug clinical trial.
* Any condition that, in the judgment of investigator, may affect trial assessment.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events during a 30 day follow-up period after each vaccination | 30 day after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Du lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Yizhou Center for Disease Control and Prevention, Yizhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: No